CLINICAL TRIAL: NCT01698853
Title: The Difference Between Central and Peripheral Arterial Blood Oxygen Saturation in Patients Undergoing Cardiac Surgery With Different Cardiopulmonary Bypass Strategy
Brief Title: Difference Between Central and Peripheral Arterial Blood Oxygen Saturation With Different CPB Strategy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 192837
Record Dates: First submitted 2012-09-25; First posted 2012-10-03 (Estimated); Last update posted 2012-10-03 (Estimated); Status verified 2012-09

CONDITIONS: Bypass Complications; Disorder of Blood Gas

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Femoro-femoral cardiopulmonary bypass with retrograde perfusion is needed for totally thoracoscopic cardiac surgery. one of the major complication of retrograde perfusion is organ hypoperfusion.

Arterial blood gas analysis can help to detect hypoperfusion or hypoxia during retrograde perfusion. However,whether the arterial oxygenation status from different parts of the body are the same in the condition of retrograde perfusion have not been studied.

The present study is aimed to determine if there is difference in the arterial oxygenation between peripheral arterial and aortic root during the period of retrograde perfusion.In addition, the impact of artificial ventilation on the difference of arterial oxygenation will also be investigated.

DETAILED DESCRIPTION:
All patients included will be assigned into two different groups according to the surgical approach,one group is named "NP" with normal perfusion,and the other is named "RP" with retrograde perfusion.

For all the patients,we will obtain 0.5ml blood from both peripheral arterial and aortic root for blood gas analysis at some specific time points.

We will focus on the differences of arterial oxygenation between peripheral arterial and aortic root at each group.At the same time,we will analyse the impact of artificial ventilation on it.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years old
* undergoing totally thoracoscopic cardiac surgery with cardiopulmonary bypass

Exclusion Criteria:

* without informed consent
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient undergoing totally thoracoscopic cardiac surgery with cardiopulmonary bypass
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2012-10; Primary Completion 2013-03 (Estimated); Study Completion 2013-05 (Estimated)

PRIMARY OUTCOMES:
The difference between peripheral arterial oxygenation and aortic root blood oxygenation | patients will be followed up during the cardiopulmonary bypass. Blood samples will be collected at 3 timepoints which is specified in the DESCRIPTION
  The three time points for blood sample collection are:1.right before clamping the aorta; 2.Three minutes after **** without ventilation;3.5 min after re-initiate mechanical ventilation.

CONTACTS AND LOCATIONS:
Overall Officials: Hailong Dong, Doctor, Study Chair — department director
Locations (1):
- Department of Anesthesiology, Xijing Hospital, Xi'an, Shaanxi, China